CLINICAL TRIAL: NCT06210542
Title: Precise Treatment of Ceftazidime-Avibactam in Patients With CRO Infections Under the Guidance of TDM and PPK Model
Status: Not yet recruiting | Type: Observational
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Lingai Pan, Associate Clinical Professor, Sichuan Provincial People's Hospital
Other Study IDs: LPan20230579
Record Dates: First submitted 2024-01-02; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: ECMO; Carbapenem-Resistant Enterobacteriaceae Infection
MeSH Terms: interventions — avibactam, ceftazidime drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: ceftazidime avibactam — Routine treatment dose for patients: the recommended intravenous dose for patients with creatinine clearance rate (eCrCL) > 50ml/min was 2.5g (2g/0.5g), once every 8 hours, and the infusion time was 2 hours.
  Patients with renal injury adjust the dosage according to eCrCL

SUMMARY:
The goal of this study is to evaluate the efficacy and safety of ceftazidime-avibactam(CAZ-AVI) in the treatment of critically ill patients with carbapenem-resistant organisms(CRO) infections (including dialysis patients and extracorporeal membrane oxygenation(ECMO) patients).

DETAILED DESCRIPTION:
This is a prospective observational multicentre study. The study is to obtain the real world data of the efficacy and safety of ceftazidime-avibactam(CAZ-AVI) in the treatment of critically ill patients with carbapenem-resistant organisms(CRO) infections (including dialysis patients and extracorporeal membrane oxygenation(ECMO) patients) by using therapeutic drug monitoring(TDM). A population-pharmacokinetic(PPK) model of CAZ-AV in these patients will be established in this study. The main question it aims to answer is the clinical success rate and microbiological success rate of CAZ-AVI based regimen in the treatment of critically ill patients with CRO infections. According to the clinical practice (symptoms, signs, imaging, culture and drug sensitivity, etc.), the doctor determines the combined regimen of CAZ-AVI, and the combined drugs are used routinely according to their instructions or clinical diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

1. 18-85 years old.
2. Hospitalized participants in ICU who did not receive Ceftazidime Avibactam treatment within 15 days before joining the study.
3. Participants with severe infection (refer to the 2022 sepsis3.0 guidelines for the definition of severe infection).
4. at least one carbapenem-resistant Gram-negative pathogen (including but not limited to carbapenem-resistant Enterobacteriaceae and / or Pseudomonas aeruginosa) was confirmed by bacterial culture in the primary infection site samples.
5. sufficient respiratory secretions, blood and peritoneal effusion can be obtained within 48 hours before the first administration for bacterial culture and drug sensitivity test.
6. intravenous injection of Ceftazidime Avibactam for more than 72 hours.
7. understand compliance with research procedures and methods, voluntarily participate in this study, and sign informed consent in writing.

Exclusion Criteria:

1. Participants are less than 18.
2. Death within 72 hours after the start of treatment.
3. Known resistance to β-lactam antibacterial drugs including cephalosporins, cephalosporin compound preparations containing β-lactamase inhibitors, or Those with a history of allergies to ceftazidime avibactam sodium for injection and its excipients.
4. No indication for treatment with ceftazidime avibactam.
5. Pregnant and lactating women.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: critically ill patients in ICU with CRO infections (including dialysis patients and ECMO patients).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Clinical success rate at the end of treatment and/or the time transfer out of ICU | the end of treatment or the time transfer out of ICU,up to 1 year.
  Clinical success includes cure or symptom improvement, which means that all symptoms and signs of patients have completely recovered or significantly improved before the end of treatment and/or the time transfer out of ICU, or imaging and other non-microbiological indicators have returned to normal. The proportion of patients with cured or improved symptoms in the total population was analyzed.
Microbiologic success rate at the end of treatment and/or the time transfer out of ICU | the end of treatment or the time transfer out of ICU,up to 1 year.
  Microbiological clearance includes clearance or presumed clearance. Clearance means that the pathogenic bacteria of the original infection have not been cultured from specimens from the original infected site after treatment; presumed clearance means that in some diseases, the disappearance of symptoms and signs makes it impossible to obtain culturable materials (such as sputum, skin pus or secretions). ), or the method of obtaining the specimen is too invasive for the recovered patient, the microbiological results are considered presumptive clearance. The microbial clearance rate is the proportion of patients who are cleared or presumed to be cleared to the total analyzed population.

SECONDARY OUTCOMES:
All-cause mortality on day 28 after drug initiation | 28 days from drug initiation
  All-cause mortality refers to the proportion of the total number of deaths caused by various causes within a certain period to the total analyzed population. It is necessary to count the number of deaths caused by various causes during this period as of the 28th day after the start of medication, using the Clopper-Pearson method. Calculate the 95% confidence interval for all-cause mortality on day 28 after drug initiation.
Infection-related mortality during hospitalization in ICU | the end of treatment or the time transfer out of ICU,up to 1 year.
  The proportion of patients who died due to infection to the total analyzed population was calculated using the Clopper-Pearson method to calculate the 95% confidence interval for infection-related mortality. It should be noted that in-hospital deaths that occur after infection symptoms improve are not considered to be related to the infection.
All-cause mortality on 90 days after drug initiation | 90 days from drug initiation
  As of the 90th day after the start of medication, the number of deaths due to various causes during this time period accounted for the proportion of the total population analyzed.
Recurrence rate of infection on day 28 after starting medication | 28 days from drug initiation
  As of the 28th day after the start of medication, the number of people whose infection was controlled and then relapsed during this time period accounted for the proportion of the total analyzed population.
Length of ICU Stay | the end of treatment or the time transfer out of ICU,up to 1 year.
  Length of stay in ICU = date of discharge from ICU - date of admission to ICU + 1.
Length of Hospital Stay (LOS) | the end of treatment or the time transfer out of ICU,up to 1 year.
  Length of stay = discharge date - admission date + 1.
Time from ceftazidime-avibactam treatment initiation to symptom improvement | the end of treatment or the time transfer out of ICU,up to 1 year.
  As an indicator of time event type, the clinical outcome of the patients was marked as the end event of symptom improvement, and the patients who did not achieve symptom improvement at the observation deadline were marked as deletion. The median value and 95% confidence interval were estimated by Kaplan-Meier method.